CLINICAL TRIAL: NCT00733772
Title: The Effects of Flaxseed Supplement on Cardio-metabolic Risk Factors in Patients With Metabolic Syndrome
Brief Title: Flaxseed Intervention on Metabolic Syndrome
Acronym: FIMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSCX1-YW-02
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Metabolic Syndrome X
Keywords: flaxseed; lignans; alpha-Linolenic Acid; LDL Cholesterol
MeSH Terms: conditions — Metabolic Syndrome | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): healthy lifestyle counseling + 30 grams/day supplement of Flaxseed
  Interventions: Dietary Supplement: flaxseed; Behavioral: Health lifestyle counseling
- B (Sham Comparator): TLC diet
  Interventions: Behavioral: Health lifestyle counseling

INTERVENTIONS:
Dietary Supplement: flaxseed — 30 grams/day of flaxseed for 12 weeks
  Arms: A
Behavioral: Health lifestyle counseling — Health lifestyle counseling accroding to AHA reccommendation
  Other Names: Health lifestyle counseling accroding to AHA reccommendation

SUMMARY:
The purpose of this study is to determine whether daily supplement of 30 grams flaxseed is effective in the treatment of metabolic syndrome (MetS).

DETAILED DESCRIPTION:
Metabolic syndrome (MetS), a constellation of metabolic abnormalities including central obesity, dyslipidemia, elevated blood pressure and hyperglycemia, is associated with the development of type 2 diabetes and CVD. It has become one of the major public health challenges in China due to rapidly nutrition transition and the nature of obesity epidemic. Treatment of MetS in China is very important for the prevention of the epidemic of its consequences (such as CVD and type 2 diabetes).

Compelling evidence from recent human studies has demonstrated that diet and lifestyle modifications are effective means in MetS management. Flaxseed is a complex food source containing high amounts of alpha-linolenic acid (ALA) - an omega-3 fatty acid - as well as fiber, lignan precursors and other substances that may have an impact on our health. Therefore, the aim of this study is to investigate the effect of flaxseed supplementation on the management of MetS in adult Chinese men and women in a randomized, controlled clinical trial. A total of 200 participants with MetS (defined by NCEP-ATPⅢ criteria) will be randomly assigned to a flaxseed-supplemented diet (30 grams/day) or an isocaloric control diet for 12 weeks. Effects of flaxseed supplementation will be evaluated by measuring metabolic profile (BMI, blood pressure, total cholesterol, triglyceride, LDL-C and HDL-C, fasting glucose and insulin, HbA1C), inflammatory markers (CRP and IL-6), markers of endothelial function (E-selectin, ICAM-1 and VCAM-1), and fatty acid profile.

ELIGIBILITY:
Inclusion Criteria:

* with metabolic syndrome Metabolic syndrome was defined based upon the updated National Cholesterol Education Program Adult Treatment Panel III criteria for Asian-Americans as presenting at least 3 of the following components: 1) waist circumference ≥ 90 cm for men or ≥ 80 cm for women; 2) triglycerides ≥1.7mmol/l; 3) HDL cholesterol <1.03 for men or <1.30 for women; 4) blood pressure ≥130/85 mmHg, or current use of antihypertentive medications; 5) fasting glucose ≥5.6mmol/l or previously diagnosed type 2 diabetes or on oral antidiabetic agents or insulin. - Being able to comply with the specified feeding conditions
* Being able to eat flaxseeds
* Being between the ages of 35 and 60 years

Exclusion Criteria:

* Pregnancy or lactation
* Use of insulin
* Severe kidney disease
* Cardiovascular diseases, stroke, cancer and psychological disorders
* Flaxseed allergies or frequently eating flaxseeds or sesame (>90 grams/week)
* Drug or alcohol abuse.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome status | 12 weeks

SECONDARY OUTCOMES:
Total cholesterol, triglyceride, HDL-C,LDL-c, fasting glucose and insulin, HbA1C, blood pressure, CRP, IL-6, adiponectin, RBP-4, E-selectin, ICAM-1, VCAM-1, and fatty acid profiles of red blood cells. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, MD, PhD, Principal Investigator — Institute for Nutritional Sciences, Chinese Academy of Sciences
Locations (1):
- Institute for Nutritional Sciences, Chinese Academy of Sciences, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu H, Pan A, Yu Z, Qi Q, Lu L, Zhang G, Yu D, Zong G, Zhou Y, Chen X, Tang L, Feng Y, Zhou H, Chen X, Li H, Demark-Wahnefried W, Hu FB, Lin X. Lifestyle counseling and supplementation with flaxseed or walnuts influence the management of metabolic syndrome. J Nutr. 2010 Nov;140(11):1937-42. doi: 10.3945/jn.110.126300. Epub 2010 Sep 8. PMID 20826632